CLINICAL TRIAL: NCT03732937
Title: Estimation of Gestational Age by Transcerebellar Diameter in Normal and Abnormal Pregnancy States
Brief Title: Estimation of Gestational Age by TCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Lecturer, Researcher , National Research centre and Consultant of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: cerebellum
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Gestational Age and Weight Conditions
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Pregnant ladies with no medical disorders from 16 weeks till term
  Interventions: Diagnostic Test: Ultrasonography
- case group: Pregnant ladies with medical disorders from 16 weeks till term
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Ultrasonography with biometry and TCD measurement

SUMMARY:
- Different parameters are used to estimate gestational age AC, HC , BPD and FL

DETAILED DESCRIPTION:
-TCD is one of the parameters ,here we are testing its accuracy in calculating GA

ELIGIBILITY:
Inclusion Criteria:

* pregnant ladies with GA between 16 - 40 weeks

Exclusion Criteria:

* pregnant ladies with GA less than 16 weeks

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females
Study Population: pregnant ladies with GA between 16 - 40 weeks
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-20 (Estimated)

PRIMARY OUTCOMES:
The number of participants who will be exactly dated by TCD in comparison to LMP | within 4 months
  The number of participants who will be exactly dated by TCD in comparison to LMP in weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt